CLINICAL TRIAL: NCT07005856
Title: The Immediate Effects of Soft Tissue Mobilization on Shoulder Mobility, Pain, Scapular Kinematics and Muscle Activation and Muscle Stiffness in Symptomatic Overhead Athletes With Posterior Shoulder Tightness
Brief Title: The Immediate Effects of Soft Tissue Mobilization on Posterior Shoulder Tightness in Overhead Athletes With Subacromial Pain Syndrome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Yang Ming Chiao Tung University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: NYCU111191AF
Record Dates: First submitted 2025-04-14; First posted 2025-06-05 (Actual); Last update posted 2025-06-05 (Actual); Status verified 2024-05

CONDITIONS: Posterior Shoulder Tightness; Subacromial Impingement Syndrome
Keywords: Posterior shoulder tightness; subacromial impingement
MeSH Terms: conditions — Shoulder Impingement Syndrome | interventions — Diathermy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Soft tissue mobilization group (Experimental)
  Interventions: Other: Soft tissue mobilization
- Stretching group (Experimental)
  Interventions: Other: Stretching
- Hot pack group (Active Comparator)
  Interventions: Other: Hot pack

INTERVENTIONS:
Other: Soft tissue mobilization — Soft tissue mobilization: mobilization participants' soft tissue by using hands
  Arms: Soft tissue mobilization group
Other: Stretching — Stretching: help patients do the movement that they're limited to stretch their soft tissue
  Arms: Stretching group
Other: Hot pack — Add an hot pack on participants' shoulder
  Other Names: heat therapy
  Arms: Hot pack group

SUMMARY:
The aim of this study is to investigate the immediate effects of soft tissue mobilization on shoulder mobility, pain, scapular kinematics and muscle activation and muscle Stiffness in symptomatic overhead athletes with posterior shoulder tightness.

ELIGIBILITY:
Inclusion Criteria:

* Amateur overhead athletes aged 18-50 years.
* Participation in overhead sports training for more than 4 hours per week.
* Playing experience of more than 3 years.
* Shoulder range of motion deficits: internal rotation range of motion (ROM) on the affected side is at least 10 degrees less than the unaffected side, and total rotational ROM (internal rotation + external rotation) is at least 5 degrees less than the unaffected side, or horizontal adduction ROM is at least 10 degrees less than the unaffected side.
* Patients with subacromial pain syndrome: diagnosis requires at least 3 out of 5 positive test results (Hawkins-Kennedy impingement test, Neer impingement test, Empty Can test, Painful Arc test, and External Rotation Resistance test).

Exclusion Criteria:

* Negative result on the kinetic medial rotation test.
* History of shoulder fracture, dislocation, or upper limb injury requiring surgery within the past 6 months.
* Inability to complete the experiment due to personal factors.
* Shoulder pain intensity greater than 7 points on the Visual Analog Scale (VAS).
* History of direct trauma to the neck or upper limb within the past month. Shoulder pain and neurological symptoms originating from the cervical spine. Contraindications to soft tissue mobilization, such as open wounds in the treatment area, skin cancer, localized infection, severe edema, vascular disorders, or acute muscle tears in the treatment area

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 54 (Actual)
Dates: Start 2024-05-15 (Actual); Primary Completion 2025-01-15 (Actual); Study Completion 2025-01-15 (Actual)

PRIMARY OUTCOMES:
Shoulder average pain intensity | Immediately after the single session
  Pain is measured with Visual Analogue scale (VAS) Score range from 0 to 10. Scoring of 0 represents no pain and scoring of 10 represents pain as bad as it could possibly be.
Shoulder passive range of motion (measured with goniometer) | Immediately after the single session
  Shoulder external rotation, internal rotation, horizontal adduction range of motion in shoulder flexion 90 degrees
Shoulder active range of motion (measured with goniometer) | Immediately after the single session
  Shoulder external rotation, internal rotation, horizontal adduction range of motion in shoulder flexion 90 degrees
Perceived improvement | Immediately after the single session
  Perceived improvement was assessed through the GROC scale. Global Rating of Change (GROC) scale was used to assess the participant's perceived improvement. The scale ranges from -7 to +7, where -7 indicates a very great deal worse, 0 indicates no change, and +7 indicates a very great deal better. Higher scores reflect greater perceived improvement.
Shoulder muscle stiffness | Immediately after the single session
  Mean dynamic muscle stiffness (N/m) of shoulder posterior muscles (deltoid, infraspinatus, teres minor) measured by MyotonPRO

SECONDARY OUTCOMES:
Surface electromyography (TeleMyo2400T G2, Noraxon USA Inc., Scottsdale, AZ, USA) | Immediately after the single session
  Muscle activation of infraspinatus, upper trapezius, lower trapezius and serratus anterior during shoulder elevation task in scapular plane and saggital plane
Scapular kinematics (degrees) during shoulder elevation measured by VIPER™ system | Immediately after the single session
  Scapular upward rotation, posterior tilt, and external rotation angles (in degrees) were recorded during shoulder elevation in the scapular and sagittal planes using the VIPER™ electromagnetic tracking system. Data were collected at 30°, 60°, 90°, and 120° of humeral elevation, and reported as mean values for each angle.

CONTACTS AND LOCATIONS:
Locations (1):
- National Yang Ming Chiao Tung University, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: Undecided